CLINICAL TRIAL: NCT01769547
Title: A Phase II Study of Single-agent DOVitinib in Advanced Malignant PlEural Mesothelioma Which Has Progressed Following Prior Platinum-Antifolate Chemotherapy
Acronym: DOVE-M
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Stage 1 accrual completed. Study did not proceed to Stage 2 accrual.
Sponsor: Ontario Clinical Oncology Group (OCOG) (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OCOG-2012-DOVE-M
Record Dates: First submitted 2013-01-09; First posted 2013-01-16 (Estimated); Last update posted 2015-09-17 (Estimated); Status verified 2015-09

CONDITIONS: Advanced Malignant Pleural Mesothelioma; MPM
MeSH Terms: interventions — 4-amino-5-fluoro-3-(5-(4-methylpiperazin-1-yl)-1H-benzimidazol-2-yl)quinolin-2(1H)-one

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Dovitinib (Experimental): Dovitinib 500 mg PO OD (5 days on, 2 days off); Each cycle = 28 days
  Interventions: Drug: Dovitinib

INTERVENTIONS:
Drug: Dovitinib — Treatment continued until Disease Progression, Toxicity, or patient withdrawal.
  Other Names: TKI258; RTK Inhibitor

SUMMARY:
This is a single-arm, open label, two stage, phase II study of dovitinib in patients with advanced Malignant Pleural Mesothelioma (MPM). The primary purpose of this study is to evaluate the potential efficacy of dovitinib in the second- or third-line treatment of MPM using progression free survival (PFS).

ELIGIBILITY:
Inclusion Criteria:

* Advanced incurable histologically confirmed malignant pleural mesothelioma that has progressed following prior administration of platinum-antifolate based chemotherapy.
* Measurable disease by RECIST 1.1. For those patients with only pleural rind, measurable disease will be determined using modified RECIST criteria.
* Availability of archival tissue.

Exclusion Criteria:

* Less than 18 years of age.
* ECOG performance status > 2.
* Received > two lines of systemic therapy.
* Patients who have received the last administration of an anticancer monoclonal antibody, immunotherapy, hormonal therapy, or chemotherapy (except nitrosureas and mitomycin-C) ≤ 4 weeks prior to starting study drug or who have not recovered from the side effects of such therapy.
* Patients who have received the last administration of nitrosureas or mitomycin-C ≤ 6 weeks prior to starting study drug, or who have not recovered from the side effects of such therapy.
* Patients who have received radiotherapy ≤ 4 weeks prior to starting the study drug or who have not recovered from radiotherapy-related toxicities (note: palliative radiotherapy for bone lesions ≤ 2 weeks prior to starting study drug is allowed).
* Patients who have undergone major surgery (e.g., intra-thoracic, intra-abdominal, intra-pelvic) ≤ 4 weeks prior to starting study treatment or who have not recovered from side effects of such surgery.
* Prior use of angiogenesis inhibitors.
* Patients with another primary malignancy within 3 years prior to starting study treatment, with the exception of adequately treated cancer such as basal cell carcinoma, squamous cell carcinoma, or non-melanomatous skin cancer or in-situ carcinoma of the uterine cervix. (Exception, patients with localized prostate cancer treated within the last 2 years and currently on hormonal therapy).
* Patients with a history of pulmonary embolism (PE), or untreated deep venous thrombosis (DVT) ≤ 6 months prior to starting study drug.
* Cirrhosis of the liver or known hepatitis B or C infection that is either acute or is considered chronic because the virus did not become undetectable:

  1. Hepatitis C Virus (HCV) infection: acute or chronic infection as depicted by a positive HCV RNA testing (note: in a patient with known anti-HCV but with a negative test for HCV RNA, re-testing for HCV RNA 4-6 months later is requested to confirm the resolution of HCV infection)
  2. Hepatitis B Virus (HBV) infection: acute infection (HBsAg+ with or without HBeAg+ or detectable serum HBV DNA), HBV carriers as evidence by ongoing presence of HBsAg and detectable serum HBV DNA levels
* Known diagnosis of human immunodeficiency virus (HIV) infection (HIV testing is not mandatory).
* Patients who are currently receiving antiplatelet therapy of prasugrel or clopidogrel, or full dose anticoagulation treatment with therapeutic doses of warfarin. However, treatment with low doses of warfarin (e.g., ≤ 2 mg/day) or locally accepted low doses of acetylsalicylic acid (up to 100 mg daily) to prevent cardiovascular events or strokes is allowed. Required use of therapeutic doses of coumarin-derivative anticoagulants such as warfarin, although doses of up to 2mg daily are permitted for prophylaxis of thrombosis. Note: Low molecular weight heparin is permitted provided the patient's PT INR is < 1.5.
* Urine dipstick reading: Positive for proteinuria or, if documentation of +1 results for protein on dipstick reading, then total urinary protein >500 mg and measured creatinine clearance <50 mL/min/1.73m2 from a 24 hour urine collection.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to dovitinib.
* Taking medications that are potent CYP3A4 inducers or inhibitors (dovitinib is metabolized primarily by the CYP3A4 liver enzyme, every effort should be made to switch patients taking such agents or substances to other medications).
* History of cardiac dysfunction with an ECHO or MUGA scan outside the institutional range of normal for patients with impaired cardiac function or clinically significant cardiac disease, including any of the following:

  1. History or presence of serious uncontrolled ventricular arrhythmias
  2. Clinically significant resting bradycardia
  3. LVEF assessed by either 2-D echocardiogram (ECHO) < 50% or lower limit of normal (whichever is the higher), or 2-D multiple gated acquisition scan (MUGA) < 45% or lower limit of normal (whichever is the higher)
  4. Any of the following within 6 months prior to starting study drug: myocardial infarction (MI), severe/unstable angina, coronary artery bypass graft (CABG), congestive heart failure (CHF), cerebrovascular accident (CVA), transient ischemic Attack (TIA)
  5. Uncontrolled hypertension defined by a SBP ≥ 160 mm Hg and/or DBP ≥ 100 mm Hg, with or without anti-hypertensive medication(s). Initiation or adjustment of antihypertensive medication(s) is allowed prior to study entry
* Pre-existing condition (e.g., gastrointestinal tract disease), resulting in an inability to take oral medication or a requirement for IV alimentation, prior surgical procedures affecting absorption, or active peptic ulcer disease that impairs the ability to swallow and retain dovitinib tablets.
* Pre-existing thyroid abnormality with an inability to maintain thyroid function in the normal range with medication.
* Patients with any of the following conditions:

  1. Clinically significant pulmonary or GI bleeding of greater than 30 cc in the preceding 3 months
  2. Serious or non-healing wound, ulcer, or bone fracture,
  3. History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 28 days of treatment.
* Patients with brain metastases.
* Other concurrent severe and/or uncontrolled concomitant medical conditions (e.g. active or uncontrolled infection, uncontrolled diabetes) that could cause unacceptable safety risks or compromise compliance with the protocol.
* Any abnormal organ and marrow function as defined below:

  1. Leukocytes <3,000/microL
  2. Absolute neutrophil count <1,500/microL
  3. Platelets <100,000/microL
  4. Total bilirubin >1.5X institutional upper limit of normal (ULN)
  5. AST(SGOT) / ALT(SGPT) >2.5X institutional ULN
  6. Amylase/lipase outside normal institutional limits
  7. Serum creatinine >1.5X ULN or Creatinine clearance <60mL/min/1.73 m2 for patients with creatinine levels above institutional normal
* Pregnant or lactating women.
* Women of child-bearing potential, who are biologically able to conceive, not employing two forms of highly effective contraception.

Note: Highly effective contraception (e.g. male condom with spermicide, diaphragm with spermicide, intra-uterine device) must be used by both sexes (female patients and their male partners) during the study and 30 days after the end of study treatment. Contraceptives that are affected by cytochrome P450 interactions (e.g. oral, implantable, injectable, or intrauterine hormonal contraceptives) are not considered effective for this study. Women of child-bearing potential, defined as sexually mature women who have not undergone a hysterectomy or who have not been naturally postmenopausal for at least 12 consecutive months (i.e., who has had menses any time in the preceding 12 consecutive months), must have a negative serum pregnancy test ≤ 14 days prior to starting study drug.

* Fertile males not willing to use contraception. Note: Fertile males must use condom with spermicide. Highly effective contraception (e.g. male condom with spermicide, diaphragm with spermicide, intra-uterine device) must be used by both sexes (male patients and their female partners) during the study and 30 days after the end of study treatment.
* Psychiatric illness/social situations that would limit compliance with study requirements.
* Receiving any other investigational agent(s).
* Patients unwilling or unable to comply with the protocol.
* Inability to understand or unable to provide written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2013-03; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | PFS measured from the time from the first date of treatment with dovitinib until the date of disease progression or date of death or last contact. Assessments every 8 weeks for disease progression for up to 2.5 years.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Response measured from the time from the first date of treatment with dovitinib. Patients should be re-evaluated for response every 8 weeks for up to 2.5 years
  ORR using the modified RECIST criteria for MPM. This is defined as the number of patients with a complete or partial response divided by the number of patients who receive at least one dose of dovitinib.
Stable disease rate/disease control rate (ORR + SD) | Stable disease measured from the time from the first date of treatment with dovitinib until the criteria for disease progression are met. Assessments every 8 weeks for disease progression for up to 2.5 years
  ORR + SD is defined as the number of patients with an objective response or stable disease using the modified RECIST criteria for MPM, divided by the number of patients who receive at least one dose of dovitinib
Duration of response / stable disease | Duration of overall response measured from the time measurement criteria are met for CR or PR until the first date that recurrent or progressive disease is objectively documented. Assessments every 8 weeks for disease progression for up to 2.5 years.
  The duration of overall CR measured from the time measurement criteria are first met for CR until the first date that recurrent disease is objectively documented.
Overall survival (OS) | OS measured from the time from the first date of treatment with dovitinib to the date of death or last contact. Patients will be followed up for survival for up to 1 year after disease progression.
Biomarker assessments using tissue and plasma samples, and imaging. | Archival tissue sample at Baseline; Plasma samples at Baseline, Cycle 1 Week 2, Cycle 2 Week 1, Cycle 3 Week 1; Chest MRI at Baseline and Day 15.
  Biomarkers analysis will include analysis of archival tissue and plasma sample (wherever safely possible). In addition, pharmacodynamic effects will be measured by diffusion weighted MRI.
Safety and tolerability | From the time from the first date of treatment with dovitinib to the date the patient completes the study; patients will be followed up for survival for up to 1 year after disease progression.
  All patients will be evaluated for toxicity. Frequency and severity of adverse events will be tabulated using counts and proportions detailing frequently occurring, serious and severe events of interest.

CONTACTS AND LOCATIONS:
Overall Officials: Scott Laurie, MD, Principal Investigator — Ottawa General Hospital Cancer Centre; Mark Levine, MD, Study Director — Ontario Clinical Oncology Group (OCOG)
Locations (5):
- Canada (5):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Northeast Cancer Centre, Health Sciences North, Greater Sudbury, Ontario
  - Juravinski Cancer Centre, Hamilton, Ontario
  - Ottawa General Hospital Cancer Centre, Ottawa, Ontario
  - Princess Margaret Hospital, Toronto, Ontario

REFERENCES:
- [Derived] Laurie SA, Hao D, Leighl NB, Goffin J, Khomani A, Gupta A, Addison CL, Bane A, Seely J, Filion ML, Pond GR, Levine MN. A phase II trial of dovitinib in previously-treated advanced pleural mesothelioma: The Ontario Clinical Oncology Group. Lung Cancer. 2017 Feb;104:65-69. doi: 10.1016/j.lungcan.2016.12.004. Epub 2016 Dec 15. PMID 28213002